CLINICAL TRIAL: NCT03832673
Title: PECULIAR: An Open Label, Monocenter, Single-arm, Phase 2 Study of Neoadjuvant Pembrolizumab and Epacadostat, Preceding Radical Cystectomy, for Patients With Muscle-invasive Bladder Cancer.
Brief Title: Pembrolizumab-Epacadostat Combination to Treat Muscle-invasive Bladder UrotheLIAl canceR: PECULIAR Study
Acronym: PECULIAR
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Regolatory National Agency (AIFA) not approved
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NT
Record Dates: First submitted 2019-01-31; First posted 2019-02-06 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Muscle-invasive Bladder Cancer
Keywords: bladder; cancer
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab; epacadostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab + Epacadostat (Experimental): Pembrolizumab 200 mg IV every 3 weeks (for 3 cycles) Epacadostat 300 mg (BID) orally continuously every 28 days (for 3 cycles)
  Interventions: Drug: Pembrolizumab; Drug: Epacadostat

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg IV every 3 weeks (for 3 cycles)
  Other Names: KEYTRUDA
Drug: Epacadostat — Epacadostat 300 mg (BID) orally continuously every 28 days (for 3 cycles)
  Other Names: previously INCB24360

SUMMARY:
An open label, monocenter, single-arm, phase 2 study of neoadjuvant pembrolizumab and epacadostat, preceding radical cystectomy, for patients with muscle-invasive bladder cancer.

DETAILED DESCRIPTION:
An open label, monocenter, single-arm, phase 2 study

ELIGIBILITY:
Inclusion Criteria:

1. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial
2. Male/female participants who are at least 18 years of age will be enrolled in this study.
3. A male participant must agree to use a contraception during the treatment period and for at least [120 days, corresponding to time needed to eliminate any study treatments) plus an additional 120 days (a spermatogenesis cycle) for study treatments with evidence of genotoxicity at any dose] after the last dose of study treatment and refrain from donating sperm during this period.
4. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: a.) Not a woman of childbearing potential (WOCBP) or b.) A WOCBP who agrees to follow the contraceptive during the treatment period and for at least [120 days (corresponding to time needed to eliminate any study treatments) plus 30 days (a menstruation cycle) for study treatments with risk of genotoxicity] after the last dose of study treatment.
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
6. Have adequate organ function as defined in the following table Specimens must be collected within 10 days prior to the start of study treatment.
7. Histopathologically confirmed transitional cell carcinoma. Patients with mixed histologies are required to have a dominant (i.e. 50% at least) transitional cell pattern.
8. Fit and planned for cystectomy (according to local guidelines).
9. Clinical stage T2-T3a confirmed by TURB
10. N0 M0 disease by CT (or MRI) + PET/CT (within 4 weeks of initial study treatment by RECIST v1.1).

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137, IDO1).
3. Has received prior systemic anti-cancer therapy including investigational agents.
4. Has received prior radiotherapy on the bladder tumor.
5. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
6. Is currently participating in or has participated in a study of an investigational agent within 4 weeks prior to the first dose of study treatment.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.

   Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded. Participants with low-risk early stage prostate cancer defined as follows are not excluded; Stage T1c or T2a with a Gleason score ≤ 6 and prostatic-specific antigen (PSA) < 10 ng/mL either treated with definitive intent or untreated in active surveillance that has been stable for the past year prior to study allocation.
9. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a known history of Human Immunodeficiency Virus (HIV).
14. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
15. Has a known history of active TB (Bacillus Tuberculosis).
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Pregnant or breastfeeding.
19. Inability to swallow tablets or capsules

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) | 12 months
  To assess whether pembrolizumab and epacadostat combination results in pathological complete response rates (herein referred to as either "pT0" or "pCR")

SECONDARY OUTCOMES:
Responses to treatment | 12 months
  To evaluate radiological response on those patients with measurable disease (at baseline). Response (CR and PR) after 3 cycles of treatment with the study drug.
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability). | 12 months
  incidence, nature and severity of all-cause and treatment-related adverse events (AE), graded with the Common Terminology Criteria for Adverse Events (CTCAE).

OTHER OUTCOMES:
PD-L1 expression and IDO1 expression | 12 months
  identify potential biomarkers that could be used for correlation with response and outcome in this setting of bladder cancer patients as well as more advanced settings in this indication.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Necchi, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale Tumori-Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellmunt J, de Wit R, Vaughn DJ, Fradet Y, Lee JL, Fong L, Vogelzang NJ, Climent MA, Petrylak DP, Choueiri TK, Necchi A, Gerritsen W, Gurney H, Quinn DI, Culine S, Sternberg CN, Mai Y, Poehlein CH, Perini RF, Bajorin DF; KEYNOTE-045 Investigators. Pembrolizumab as Second-Line Therapy for Advanced Urothelial Carcinoma. N Engl J Med. 2017 Mar 16;376(11):1015-1026. doi: 10.1056/NEJMoa1613683. Epub 2017 Feb 17. PMID 28212060
- [Background] Disis ML. Immune regulation of cancer. J Clin Oncol. 2010 Oct 10;28(29):4531-8. doi: 10.1200/JCO.2009.27.2146. Epub 2010 Jun 1. PMID 20516428
- [Background] Dudley ME, Wunderlich JR, Yang JC, Sherry RM, Topalian SL, Restifo NP, Royal RE, Kammula U, White DE, Mavroukakis SA, Rogers LJ, Gracia GJ, Jones SA, Mangiameli DP, Pelletier MM, Gea-Banacloche J, Robinson MR, Berman DM, Filie AC, Abati A, Rosenberg SA. Adoptive cell transfer therapy following non-myeloablative but lymphodepleting chemotherapy for the treatment of patients with refractory metastatic melanoma. J Clin Oncol. 2005 Apr 1;23(10):2346-57. doi: 10.1200/JCO.2005.00.240. PMID 15800326
- [Background] Hunder NN, Wallen H, Cao J, Hendricks DW, Reilly JZ, Rodmyre R, Jungbluth A, Gnjatic S, Thompson JA, Yee C. Treatment of metastatic melanoma with autologous CD4+ T cells against NY-ESO-1. N Engl J Med. 2008 Jun 19;358(25):2698-703. doi: 10.1056/NEJMoa0800251. PMID 18565862
- [Background] Greenwald RJ, Freeman GJ, Sharpe AH. The B7 family revisited. Annu Rev Immunol. 2005;23:515-48. doi: 10.1146/annurev.immunol.23.021704.115611. PMID 15771580
- [Background] Okazaki T, Maeda A, Nishimura H, Kurosaki T, Honjo T. PD-1 immunoreceptor inhibits B cell receptor-mediated signaling by recruiting src homology 2-domain-containing tyrosine phosphatase 2 to phosphotyrosine. Proc Natl Acad Sci U S A. 2001 Nov 20;98(24):13866-71. doi: 10.1073/pnas.231486598. Epub 2001 Nov 6. PMID 11698646
- [Background] Zhang X, Schwartz JC, Guo X, Bhatia S, Cao E, Lorenz M, Cammer M, Chen L, Zhang ZY, Edidin MA, Nathenson SG, Almo SC. Structural and functional analysis of the costimulatory receptor programmed death-1. Immunity. 2004 Mar;20(3):337-47. doi: 10.1016/s1074-7613(04)00051-2. PMID 15030777
- [Background] Chemnitz JM, Parry RV, Nichols KE, June CH, Riley JL. SHP-1 and SHP-2 associate with immunoreceptor tyrosine-based switch motif of programmed death 1 upon primary human T cell stimulation, but only receptor ligation prevents T cell activation. J Immunol. 2004 Jul 15;173(2):945-54. doi: 10.4049/jimmunol.173.2.945. PMID 15240681
- [Background] Sheppard KA, Fitz LJ, Lee JM, Benander C, George JA, Wooters J, Qiu Y, Jussif JM, Carter LL, Wood CR, Chaudhary D. PD-1 inhibits T-cell receptor induced phosphorylation of the ZAP70/CD3zeta signalosome and downstream signaling to PKCtheta. FEBS Lett. 2004 Sep 10;574(1-3):37-41. doi: 10.1016/j.febslet.2004.07.083. PMID 15358536
- [Background] Riley JL. PD-1 signaling in primary T cells. Immunol Rev. 2009 May;229(1):114-25. doi: 10.1111/j.1600-065X.2009.00767.x. PMID 19426218
- [Background] Parry RV, Chemnitz JM, Frauwirth KA, Lanfranco AR, Braunstein I, Kobayashi SV, Linsley PS, Thompson CB, Riley JL. CTLA-4 and PD-1 receptors inhibit T-cell activation by distinct mechanisms. Mol Cell Biol. 2005 Nov;25(21):9543-53. doi: 10.1128/MCB.25.21.9543-9553.2005. PMID 16227604
- [Background] Francisco LM, Sage PT, Sharpe AH. The PD-1 pathway in tolerance and autoimmunity. Immunol Rev. 2010 Jul;236:219-42. doi: 10.1111/j.1600-065X.2010.00923.x. PMID 20636820
- [Background] Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, Lin NU, Litiere S, Dancey J, Chen A, Hodi FS, Therasse P, Hoekstra OS, Shankar LK, Wolchok JD, Ballinger M, Caramella C, de Vries EGE; RECIST working group. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol. 2017 Mar;18(3):e143-e152. doi: 10.1016/S1470-2045(17)30074-8. Epub 2017 Mar 2. PMID 28271869
- [Background] Necchi A, Rink M, Giannatempo P, Raggi D, Xylinas E. Immunotherapy for metastatic urothelial carcinoma: status quo and the future. Curr Opin Urol. 2018 Jan;28(1):1-7. doi: 10.1097/MOU.0000000000000457. PMID 29028766
- [Background] Mitchell TC, Hamid O, Smith DC, Bauer TM, Wasser JS, Olszanski AJ, Luke JJ, Balmanoukian AS, Schmidt EV, Zhao Y, Gong X, Maleski J, Leopold L, Gajewski TF. Epacadostat Plus Pembrolizumab in Patients With Advanced Solid Tumors: Phase I Results From a Multicenter, Open-Label Phase I/II Trial (ECHO-202/KEYNOTE-037). J Clin Oncol. 2018 Nov 10;36(32):3223-3230. doi: 10.1200/JCO.2018.78.9602. Epub 2018 Sep 28. PMID 30265610
- [Background] Necchi A, Anichini A, Raggi D, Briganti A, Massa S, Luciano R, Colecchia M, Giannatempo P, Mortarini R, Bianchi M, Fare E, Monopoli F, Colombo R, Gallina A, Salonia A, Messina A, Ali SM, Madison R, Ross JS, Chung JH, Salvioni R, Mariani L, Montorsi F. Pembrolizumab as Neoadjuvant Therapy Before Radical Cystectomy in Patients With Muscle-Invasive Urothelial Bladder Carcinoma (PURE-01): An Open-Label, Single-Arm, Phase II Study. J Clin Oncol. 2018 Dec 1;36(34):3353-3360. doi: 10.1200/JCO.18.01148. Epub 2018 Oct 20. PMID 30343614